CLINICAL TRIAL: NCT02881762
Title: A Pilot Study to Evaluate Anti-Hepatitis C Virus Effect of Maraviroc in Patients Co-infected With Human Immunodeficiency Virus (HIV) and Hepatitis C
Brief Title: Maraviroc Efficacy for Hepatitis C
Acronym: MAVERIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Lydia Tang, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP-00070324
Record Dates: First submitted 2016-08-10; First posted 2016-08-29 (Estimated); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2023-10

CONDITIONS: Hepatitis C; Human Immunodeficiency Virus
Keywords: hepatitis C virus (HCV); Maraviroc; Human immunodeficiency virus (HCV)
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate start maraviroc (Active Comparator): To start maraviroc immediately after randomization.
  Interventions: Drug: Maraviroc
- Delayed start maraviroc (Active Comparator): To start maraviroc 8 weeks after enrollment.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Participants will receive 4 weeks of maraviroc (dosing based on concomitant HIV antiretroviral regimen). Serial measurements of HCV viral load will be obtained before, during, and after maraviroc exposure. Study duration will be approximately 12 to 16 weeks.
  Other Names: Selzentry

SUMMARY:
This is a single-site, longitudinal, open-label, interventional study for evaluating the effect of maraviroc on hepatitis C viral levels in patients infected with both hepatitis C and human immunodeficiency virus (HIV) and taking antiretroviral therapy for HIV.

DETAILED DESCRIPTION:
Recently, in-vitro studies (experiments performed in a laboratory, not on a person) have demonstrated that maraviroc, a medication that is used in human immunodeficiency (HIV) therapy, appears to have significant hepatitis C antiviral effect, comparable to sofosbuvir-a potent anti-hepatitis C medication. In this study, the investigators will evaluate the antiviral effect of maraviroc on hepatitis C virus in people infected with both hepatitis C and HIV, and whom have never been treated for hepatitis with direct antiviral agents. Participants will take maraviroc for 4 weeks in addition to their regular HIV antiretrovirals (ART). The investigators will measure the hepatitis C viral load before, during, and after the 4-week maraviroc time.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old
2. Hepatitis C-infected without plans to undergo hepatitis C treatment for duration of the study
3. Human immunodeficiency virus (HIV) infected
4. Currently receiving anti-retroviral therapy with HIV viral load <50 IU/ml for ≥ 12 months

   a. One virologic blip ≤ 400 copies/ml permissible within the 12 months
5. CD4 T cell counts > 100 cells/mm3
6. Non-cirrhotics and cirrhotics can be included
7. Willing to sign informed consent

Exclusion Criteria:

1. Age < 18
2. Unable to comply with study visits, research study visits, or is planning to relocate during the study.
3. Have any condition that the investigator considers a contraindication to study participation
4. Pregnancy or breast feeding
5. Decompensated liver disease (Child-Pugh C)
6. Imminent treatment for hepatitis C infection
7. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times the upper limits of normal
8. Concomitant use of drugs known to impact or be impacted in terms of pharmacokinetics or drug-drug interactions with either raltegravir, dolutegravir, or maraviroc. This includes:

   * Inducers of UGT1A1 (such as rifampin, phenytoin, phenobarbital rifabutin, St. John's wort)
   * Cytochrome P3A inhibitors (such as ketoconazole, itraconazole, clarithromycin, nefazodone, and telithromycin)
   * Cytochrome P3A inducers (such as rifampin, carbamazepine, phenobarbital and phenytoin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyida Tang, MBChB, Principal Investigator — Assistant Professor
Locations (1):
- Institute of Human Virology at the University of Maryland School of Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at the clinical research unit at the University of Maryland, Baltimore between June 2017 to April 2018
Groups:
- Maraviroc First, Then No Maraviroc: Participants first received maraviroc, 150mg to 600mg (dose based on concomitant HIV antiretroviral regimen) twice a day for 4 weeks. After a washout period of 4 weeks, they then received no maraviroc for 4 weeks.
- No Maraviroc First, Then Maraviroc: Participants first received no maraviroc for 4 weeks. After a washout period of 4 weeks, they then received maraviroc, 150mg to 600mg (dose based on concomitant HIV antiretroviral regimen) twice a day for 4 weeks. Participants are then seen for their last visit 4 weeks after their last dose of maraviroc.
Period: First Intervention (4 Weeks)
Arm/Group | Maraviroc First, Then No Maraviroc | No Maraviroc First, Then Maraviroc
Started | 5 | 5 (1 participants signed consent, but withdrew before day 0.)
Completed | 5 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (4 Weeks)
Arm/Group | Maraviroc First, Then No Maraviroc | No Maraviroc First, Then Maraviroc
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Maraviroc First, Then No Maraviroc | No Maraviroc First, Then Maraviroc
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Followup No Maraviroc First Only (4 Wks)
Arm/Group | Maraviroc First, Then No Maraviroc | No Maraviroc First, Then Maraviroc
Started | 5 (Completed study after intervention 3 (week 12)) | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maraviroc First, Then no Maraviroc | No Maraviroc First, Then Maraviroc | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (3.1) | 55.8 (9.7) | 56.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9
Hepatitis C viral load [Mean (Standard Deviation); unit: International Units/ml] | 1734274 (949012) | 2411068 (1093469) | 2035071 (1012880)
Alanine transaminase [Mean (Standard Deviation); unit: International Units/ml] | 39.6 (21.2) | 31.8 (2.6) | 36.1 (15.7)

OUTCOME MEASURES:

1. Primary Outcome: The Change in Hepatitis C Viral Load From Baseline to 4 Weeks of Maraviroc or No Maraviroc
Description: Hepatitis C viral load was measured before starting maraviroc, and at 4 weeks of maraviroc.
Time Frame: Baseline to 4 weeks
Population: All participants who received at least one dose of each intervention and completed all study visits were included in the final analysis
Measure: Mean (Standard Deviation); unit: International Units/ml
Groups:
- Maraviroc: Participants who received Maraviroc daily either in the first 4 weeks or during week 8 to week 12
- No Maraviroc: Participants who received No Maraviroc daily either the first 4 weeks or during weeks 8 to 12 of the study.
Arm/Group | Maraviroc | No Maraviroc
Number analyzed (Participants) | 9 | 9
International Units/ml
  HCV viral load at baseline | 2035071 (1012880) | 2027648 (1411027)
  HCV viral load at 4 weeks | 2082302 (1673228) | 1216383 (769289.8)
  Change in HCV viral load at 4 weeks | 47231 (805651.4) | -811264 (1357476)
Statistical Analysis 1: Comparison: Maraviroc vs No Maraviroc; Null hypothesis is that there is no difference in change in HCV viral load between Maraviroc and No Maraviroc; Test type: Other — Comparison of mean change analyzed with unpaired t-test for parametric data. The test was performed with a significance level of 0.05 (two-sided); p = 0.13, t-test, 2 sided

2. Secondary Outcome: Change in Hepatitis C Viral Loads From Baseline to Day 7 on Maraviroc
Description: HCV viral load was measured before starting and at 7 days of maraviroc. Among participants that received Maraviroc in the first 4 weeks, HCV viral load was measured before first dose at day 0 and at day 7. Among participants that received Maraviroc in week 8 to 12, HCV viral load measured at day 56 before taking the first dose of Maraviroc and at day 63 (week 9) of study.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: International Units/ml
Groups:
- Baseline, Pre-maraviroc: HCV viral load at day 0 (in participants that received maraviroc in the first 4 weeks of study) or day 56 (in participants that received maraviroc in weeks 8 to 12 of study).
- 7 Days of Maraviroc: HCV viral measured at day 7 (in participants that received maraviroc in the first 4 weeks of study) or week 9 (in participants that received maraviroc in weeks 8 to 12 of study).
Arm/Group | Baseline, Pre-maraviroc | 7 Days of Maraviroc
Number analyzed (Participants) | 9 | 9
International Units/ml | 2035071 (1012880) | 2138768 (1732285)
Statistical Analysis 1: Comparison: Baseline, Pre-maraviroc vs 7 Days of Maraviroc; Null hypothesis is that there is no difference in HCV viral load between baseline and 7 days of maraviroc; Test type: Other — Comparison of difference in mean analyzed with paired t-test for parametric data. The test was performed with a significance level of 0.05 (two-sided); p > 0.5, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Day 0 to end of study (week 12 for immediate start, week 16 for delayed start)
Arm/Group | Maraviroc | No Maraviroc
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc (N=9) | No Maraviroc (N=9)
Tibial plateau fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — tripped over curb and sustained fracture requiring hospitalization. Not related to study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc (N=9) | No Maraviroc (N=9)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — 1 episode
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) — 1 episode, resolved after sitting down for 10 minutes
Soft tissue injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — stepped on sharp object and hurt big toe
Bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — post phlebotomy bruise

LIMITATIONS AND CAVEATS:
Small numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT02881762/Prot_SAP_000.pdf